CLINICAL TRIAL: NCT02124915
Title: Influence of Socket Volume on Prosthesis Performance
Acronym: CAD
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Joan Sanders, Professor, University of Washington
Other Study IDs: STUDY00001507; R01HD069387 (NIH)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Lower Limb Amputation Below Knee (Injury)
Keywords: prosthetic socket; amputee
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transtibial amputees

SUMMARY:
The purpose of this study is to investigate how residual limb fluid volume, gait, prosthesis use, perceived comfort, and satisfaction with the prosthesis are affected by size of the prosthetic socket. Subjects are tested after wearing a nominal socket for 1 month and again after wearing a slightly oversized socket for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* transtibial amputee
* at least 18 months post amputation
* over 18 years of age
* capable of treadmill walking and 90 seconds of continuous standing

Exclusion Criteria:

* skin breakdown on the residual limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transtibial amputees
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Residual limb fluid volume | 1 month

SECONDARY OUTCOMES:
Activity | 1 month

OTHER OUTCOMES:
Comfort and prosthesis satisfaction | 1 month
Gait | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States